CLINICAL TRIAL: NCT04798846
Title: Spanning Plate Versus Spanning External Fixator in Fixation of Comminuted Distal Radius Fracture
Brief Title: Fixation of Comminuted Distal Radius Fracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Eslam Abdelnaby Abdelsabor, principal investigator, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh_Med_21_02_11
Record Dates: First submitted 2021-02-23; First posted 2021-03-15 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Distal Radius Fracture
Keywords: distal radius fracture
MeSH Terms: conditions — Wrist Fractures | interventions — External Fixators

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- External fixator (Active Comparator): patient treated by external fixator
  Interventions: Procedure: dorsal plating
- Dorsal plate (Active Comparator): patient treated by dorsal spanning plate
  Interventions: Procedure: dorsal plating

INTERVENTIONS:
Procedure: dorsal plating — Spanning Plate inserted dorsally below tendons Spanning External Fixator by rods inserted in distal radius and metacarpals
  Other Names: External fixator

SUMMARY:
comparison between different methods in fixation of comminuted distal radius fractures

DETAILED DESCRIPTION:
This clinical study aims at comparison of treatment outcomes of Spanning plate versus spanning External fixator in fixation of comminuted distal radius fracture.

The primary outcomes that we like to measure are pain, healing. Stiffness and range of motion .

ELIGIBILITY:
* Inclusion criteria

  * Skeletally mature patients aging 18 or more
  * Comminuted distal radius fractures Fernandez type V
* Exclusion criteria

  * Age less than 18 year or more
  * Patients with previous fracture affecting wrist joint in the same side.
  * Parients with active infection in the affected joint
  * Pathological fracture
  * Neurological disorder (epilepsy…etc) Reheumatoid

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Mayo modified wrist score | up to 6 month
  measure.grip strength

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt